CLINICAL TRIAL: NCT05776719
Title: Efficacy of Virtual Warrior Renew Therapy for Veterans Who Experienced Military Sexual Trauma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Amanda Wood, Clinical Research Psychologist, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: W81XWH-22-1-1114
Record Dates: First submitted 2023-02-23; First posted 2023-03-20 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Military Sexual Trauma (MST); Post Traumatic Stress Disorder
Keywords: group therapy; military sexual trauma; randomized clinical trial; PTSD; MST
MeSH Terms: conditions — Military Sexual Trauma; Stress Disorders, Post-Traumatic | interventions — Health

STUDY DESIGN:
Intervention Model Description: 1:1 randomization to either targeted group intervention or control group intervention; groups separated by gender
Masking Description: Study participants will be informed that they will be randomized to one of two groups but will not be informed which group is expected to perform better.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health & Wellness (Active Comparator): 8 weeks, once weekly 90 minute sessions, groups of 8-10 subjects, gender stratified
  Interventions: Behavioral: Health & Wellness
- Warrior Renew (Experimental): 8 weeks, once weekly 90 minute sessions, groups of 8-10 subjects, gender stratified
  Interventions: Behavioral: Warrior Renew

INTERVENTIONS:
Behavioral: Health & Wellness — PowerPoint slide decks will be shown via shared screen. The wellness group will be largely educational in nature and will encourage discussion, setting goals, and making healthy choices. Similar topics covered in this group have been used previously in health promotion classes.
  Arms: Health & Wellness
Behavioral: Warrior Renew — The group format includes warm-up community building exercises, psychoeducational presentation of material standardized by the use of PowerPoint slides, followed by discussion of the information and interactive exercises, and closes with exercises to improve affect management skills, such as mindfulness or guided imagery.
  Arms: Warrior Renew

SUMMARY:
Group treatments may be helpful for Veterans who have experienced military sexual trauma (MST). By doing this study, the investigators hope to learn if two different groups: Warrior Renew and Health & Wellness are effective in reducing mental health symptoms in Veterans who have experienced MST and if either is more effective than the other. Participation in this research will last about 16 weeks.

DETAILED DESCRIPTION:
This project will examine mental health treatment in a group setting for Veterans who have experienced military sexual trauma. Military sexual trauma or MST is defined as any experience of sexual assault or sexual harassment experienced during military service. Survivors of MST may develop mental health symptoms. Group treatment for survivors of MST may be helpful. This study will compare two different group treatments: 1) Warrior Renew; and 2) Health & Wellness.

By doing this study, the investigators hope to learn: 1) if one or both of the group treatments are safe and effective in reducing mental health symptoms in Veterans who have experienced MST; and 2) if there are differences based on gender that should be addressed differently in developing treatments for survivors of MST.

ELIGIBILITY:
Inclusion Criteria:

1. Has established care with VA medical or mental health provider.
2. Reports having experienced military sexual trauma.
3. Between the ages of 18 and 75.
4. Is an outpatient and is able to comply with all study procedures, including the eight weeks of group treatment and the assessment measures.
5. Positive screen on the Primary Care PTSD Screen for DSM-5 (PC-PTSD-5).
6. Able to participate in virtual group therapy via telehealth.

Exclusion Criteria:

1. Impaired decision-making capacity that in the clinical judgment of their provider would affect their ability to provide informed consent.
2. Current/active suicidal ideation as evidenced by a positive screen on the Columbia Suicide Severity Rating Scale (C-SSRS), or a suicide attempt or psychiatric hospitalization within the past year.
3. Dissociative, delusional or psychotic symptoms due to medical conditions or mental health disorders that in the clinical judgement of the PI or LSI would impede the participant's ability to participate actively in the study.
4. Current/active diagnosis of a substance use disorder or an alcohol use disorder as measured by the Alcohol Use Disorders Identification Test-Concise (AUDIT-C).
5. Unable to read English.
6. Currently receiving trauma-focused group or individual psychotherapy treatment. (Previous psychotherapy, current pharmacotherapy, peer support groups, or maintenance therapy groups or individual therapy, defined as therapeutic services that have been ongoing for at least three months and are not trauma-focused, is acceptable).
7. Concurrently enrolled in another research protocol involving a mental health intervention during this study.
8. Has had previous Warrior Renew treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The groups will be separated by sex (e.g., men's group or women's group). Participants of all identities are invited to participate and will choose their group. Dividing the groups by sex respects possible issues of discomfort and allows for gender-specific nuanced conversations.
Enrollment: 191 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
PTSD Checklist for DSM-5 (PCL-5) | Changes from baseline to end of 8-week treatment.
  The 20-item PCL-550 will be used to assess symptoms of PTSD using items consistent with the Diagnostic and Statistical Manual 5 (DSM-5, 2013) criteria for PTSD. The wording of PCL-5 items reflects both changes to existing symptoms and the addition of new symptoms in DSM-5. The PCL-5 uses a self-report Likert rating scale of 0-4 for each symptom, including the anchors of: "Not at all," "A little bit," "Moderately," "Quite a bit," and "Extremely." A score of 31-33 has been identified as the optimally efficient cutoff for a probable diagnosis of PTSD (VA National Center for PTSD, 2015).

SECONDARY OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The PHQ-9 is self-report, nine-item screening tool for depression. The tool rates the frequency of depressive symptoms based on DSM-5 criteria for major depression, asking respondents rate each item according to the following instructions, "Over the last 2 weeks how often have you been bothered by any of the following:" Items are rated via four choices: 0= not at all, 1= several days, 2 = more than half the days, and 3= nearly every day. Scores are summed with higher scores indicating higher level of psychological distress. The PHQ-9 has been shown to have a sensitivity of 88% and specificity of 88% for Major Depression, with a Cronbach alpha of .89 (Kroenke et al., 2001). It has suggested interpretations of 5-9 = mild, 10-14 = moderate, 15-19 = moderate severe, and 20-27 = severe depression.
Generalized Anxiety Disorder Assessment (GAD-7) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The GAD-7 is a 7-item self-report measure of general anxiety. Respondents rate each item according to the following instructions, "Over the last 2 weeks how often have you been bothered by any of the following:" Items are rated via four choices: 0= not at all, 1= several days, 2 = more than half the days, and 3= nearly every day. Scores are summed with higher scores indicating higher level of psychological distress. The GAD-7 has been shown to have an 89% sensitivity and a 82% specificity for identifying general anxiety disorder, based on DSM-5.
Dimensions of Anger Reactions-5 (DAR-5) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The DAR-5 is a 7-item measure of anger that contains four questions about anger response (frequency, intensity, duration, and physical antagonism), and three items related to anger functional impairment (adverse impact on social relationships, work, and health). The revised version of this measure will be used, which reduced the Likert scale responses from nine to five items with no loss of validity. The measure has shown good internal consistency, with a Cronbach's alpha of .77 for anger response and .85 for anger impairment. Test-retest reliability was .66 for anger response and .56 for anger impairment. The scale has also shown good construct validity, showing significant correlations with all seven subscales of the longer State-Trait Anger Expression Inventory (STAXI).
Internalized Shame Scale (ISS) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The ISS is a 30-item self-report measure of trait shame, comprised of a 24-item internalized shame subscale and a 6-item self-esteem sub-scale. The measure asks about different experiences of shame without actually using the word "shame", which can be triggering and difficult to admit. A score of 50 or higher is purported to represent problematic levels of shame. The measure has shown strong internal consistency and reliability on both the internalized shame and self-esteem subscales with alpha coefficients of .88 and .96, and test-retest relatability of .81 and .75 respectively.
Posttraumatic Cognitions Inventory (PTCI) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The 33-item PTCI was used to assess trauma-related thoughts and beliefs. The PTCI has three subscales: negative cognitions about the self, negative cognitions about the world, and self-blame as well as a global scale, total negative cognitions, which is the sum of the three subscales. Items are rated using a seven-point Likert-type response scale that ranges from 1 = totally disagree, to 7 = totally agree. Negative thinking scores are computed by summing the items in each subscale with higher scores indicating higher ratings of negative thinking. The PTCI has demonstrated good internal consistency, test-retest reliability, and validity.
Attitudes towards Emotional Expression Scale (AEE) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The AEE is a 20-item scale that measures the belief that the expression of emotions is a sign of weakness (weakness); the belief that emotions should be kept under control (control); the belief that other people will reject expressed emotions (social); and the tendency to keep emotions to oneself (non-expression). Respondents are asked to respond to each item on a 5-point Likert scale ranging from strongly disagree (1) to strongly agree (5) so that scores on the total scale have a possible range of 20 to 100, with higher scores indicating more negative attitudes toward emotional expression. It is reliable, single total score with alpha reliability of .93, and valid with high correlation with the Emotional Expression Questionnaire (r = .62, p<.001).
Veteran RAND 12-Item Health Survey (VR-12) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The VR-12 is a 12-item instrument primarily used to measure health related quality of life and disease burden. The instrument summarizes both physical health and mental health influences on overall quality of life. The VR-12 was derived from the Veterans RAND 36 Item Health Survey and has been used extensively with a Veteran population.
Pain, Enjoyment of Life and General Activity Scale (PEG) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The PEG is a three-item scale of pain, derived from the Brief Pain Inventory, and includes items of pain intensity (P), interference with enjoyment of life (E), and interference with general activity (G). Overall, reliability of the PEG was good (0.73 and 0.89 in two samples). Construct validity for the PEG was also good for pain-specific measures (Krebs et al., 2009).
Pain Self-Efficacy Questionnaire (PSEQ) | Changes from baseline to after 8-week treatment and at end of 16-week follow up.
  The PSEQ is a 2-item questionnaire of pain, derived from the 10-item PSEQ. The 2-item scale has shown good validity and internal consistency, and had good convergent validity (Nicholas et al., 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Amanda E Wood, PhD, Principal Investigator — VA Puget Sound Health Care System
Locations (2):
- United States (2):
  - VA Portland Health Care System, Portland, Oregon
  - VA Puget Sound Health Care System, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
As per our current IRB restrictions, no individual participant data will be available to outside researchers.